CLINICAL TRIAL: NCT05777876
Title: Early Identification of Treatment-resistant Depression and Construction and Clinical Validation of Non-invasive Transcranial Deep Brain Stimulation Precision Technology
Brief Title: Early Identification of TRD and Construction and Clinical Validation of NTBS Precision Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Collaborators: Zhejiang University (Other); Kangci Hospital of Jiaxing (Unknown); Wenzhou Seventh People's Hospital (Other Government); Lishui Second People's Hospital (Unknown); Huzhou Third People's Hospital (Other); Binjiang Institute of Zhejiang University (Unknown); Zhejiang Newways Medical Technology Co., Ltd (Unknown); Hangzhou Lingnao Technology Co., Ltd (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Other
Other Study IDs: 2023C03077
Record Dates: First submitted 2023-02-07; First posted 2023-03-21 (Actual); Last update posted 2023-03-21 (Actual); Status verified 2023-01

CONDITIONS: Treatment-Resistant Depression
Keywords: non-invasive transcranial deep brain stimulation; Temporal Interference Stimulation; depression; early recognition
MeSH Terms: conditions — Depressive Disorder, Treatment-Resistant; Depression

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (9):
- non-TRD (No Intervention): Patients with first episode or relapse of untreated depression group are treated with escitalopram for 8 weeks, and if effective, they are included in the n-TRD group. If ineffective, Venlafaxine is used for full treatment for 8 weeks; if effective, the patients are included in the non-TRD group. The subjects get clinical evaluation, blood sample collection, magnetic resonance scanning, and electrophysiological monitoring.
- TRD Target stimulation A (Experimental): Patients do not respond favorably to two antidepressants. The subjects get clinical evaluation, blood sample collection, magnetic resonance scanning, and electrophysiological monitoring. Regimen: Receiving TIS intervention with target A (Characteristic abnormal brain region targets based on data-driven exploration) for 10 times, once a day (except weekends and holidays) for 2 weeks. Stimulation（130Hz, 2mA total current intensity, each stimulation lasts for 30 minutes, 15 seconds respectively for import and exit).
  Interventions: Device: non-invasive transcranial deep brain stimulation
- TRD Target stimulation B (Experimental): Patients do not respond favorably to two antidepressants. The subjects get clinical evaluation, blood sample collection, magnetic resonance scanning, and electrophysiological monitoring. Regimen: Receiving TIS intervention with target B (Characteristic abnormal brain region targets based on data-driven exploration) for 10 times, once a day (except weekends and holidays) for 2 weeks. Stimulation（130Hz, 2mA total current intensity, each stimulation lasts for 30 minutes, 15 seconds respectively for import and exit).
  Interventions: Device: non-invasive transcranial deep brain stimulation
- TRD Target stimulation C (Experimental): Patients do not respond favorably to two antidepressants. The subjects get clinical evaluation, blood sample collection, magnetic resonance scanning, and electrophysiological monitoring. Regimen: Receiving TIS intervention with target C (Characteristic abnormal brain region targets based on data-driven exploration) for 10 times, once a day (except weekends and holidays) for 2 weeks. Stimulation（130Hz, 2mA total current intensity, each stimulation lasts for 30 minutes, 15 seconds respectively for import and exit).
  Interventions: Device: non-invasive transcranial deep brain stimulation
- TRD sham stimulation (Sham Comparator): Patients do not respond favorably to two antidepressants. The subjects get clinical evaluation, blood sample collection, magnetic resonance scanning, and electrophysiological monitoring. Regimen: sham stimulation for 10 times, once a day (except weekends and holidays) for 2 weeks. Stimulation（130Hz, 2mA total current intensity, each stimulation lasts for 30 seconds, total wearing the instrument for 30 minutes)
  Interventions: Device: Sham stimulation
- TRD closed-loop stimulation (Experimental): Patients do not respond favorably to two antidepressants. The subjects get clinical evaluation, blood sample collection, magnetic resonance scanning, and electrophysiological monitoring. Patients receive closed-loop stimulation guided by EEG phase, and the stimulation target is the effective deep brain region target verified in this study. Regimen: stimulation for 10 times, once a day (except weekends and holidays) for 2 weeks. Stimulation（130Hz, 2mA total current intensity, each stimulation lasts for 30 minutes, 15 seconds respectively for import and exit)
  Interventions: Device: non-invasive transcranial deep brain stimulation with closed-loop
- HC experimental stimulation (Experimental): The subjects get clinical evaluation, blood sample collection, magnetic resonance scanning, and electrophysiological monitoring. HC will receive TIS intervention in the exercise area for one time, the stimulation scheme adopted 20 Hz and 2mA total current intensity, and each stimulation lasted for 30 minutes (15 seconds respectively for lead-in and withdrawal)
  Interventions: Device: Motor cortex stimulation
- HC sham stimulation (Sham Comparator): The subjects get clinical evaluation, blood sample collection, magnetic resonance scanning, and electrophysiological monitoring. Electrode placement, current intensity and intervention times are consistent with those of TIS regimen. 20 Hz, 2mA total current intensityis used, but only lasted for 30 seconds, and then the current is 0 for a total of 30 minutes.
  Interventions: Device: Sham stimulation
- HC observation (No Intervention): Collect data on healthy controls without stimulation. The subjects get clinical evaluation, blood sample collection, magnetic resonance scanning, and electrophysiological monitoring.

INTERVENTIONS:
Device: non-invasive transcranial deep brain stimulation — A new non-invasive transcranial deep brain stimulation, Temporal Interference Stimulation (TIS), can focus the stimulation region specifically on the deep brain region without affecting the upper level of the target region. At present, the safety of this method has been preliminarily verified in animals and healthy people, but the brain target of TRD treatment is not clear.
  Arms: TRD Target stimulation A; TRD Target stimulation B; TRD Target stimulation C
Device: Sham stimulation — Electrodes will be placed in the same location on the head as that for the TI intervention; 30 seconds of electrical current will be delivered to the brain (compared to 30 minutes in the experimental intervention arm), therefore it is expected to elicit no changes in neural activity.
  Arms: HC sham stimulation; TRD sham stimulation
Device: Motor cortex stimulation — Receive stimulation in the motor cortex stimulation instead of deep brain.
  Arms: HC experimental stimulation
Device: non-invasive transcranial deep brain stimulation with closed-loop — Non-invasive transcranial deep brain stimulation devices based on closed-loop regulation of EEG can improve the accuracy of treatment.
  Arms: TRD closed-loop stimulation

SUMMARY:
The goal of this clinical trial is to learn about the characteristics, identify early and intervene effectively in time in Treatment-Resistant Depression. The main questions are: • TRD is difficult to identify early and lacks objective detection indicators; • Existing treatment strategies for TRD are associated with side effects and high treatment resistance; • Current non-invasive brain stimulation therapy lacks precision.

it aims to answer are: • Construct a multimodal TRD early identification model based on clinical characteristics, blood factors, functional magnetic resonance and brain electrophysiological indicators; • Develop non-invasive transcranial deep brain stimulation technology based on focused electric field; • In TRD patients, an individualized non-invasive transcranial deep electrical stimulation technology based on precise magnetic resonance targets and EEG phase guidance was constructed.

Participants will:• be collected data multiple times including clinical symptoms, peripheral biology, functional magnetic resonance, electrophysiology and other clinical data before and after the intervention; • receive non-invasive transcranial deep brain stimulation or sham stimulation of different deep brain target points; • be collected EEG data while receiving stimulation.

Researchers will • compare the biological characteristics of TRD, n-TRD patients and health controls to build early identification models and find potential spatial and temporal intervention targets dependent on TRD status; • verify the safety of non-invasive transcranial deep brain stimulation device in health controls; • compare TRD with different modes of stimulation to find the best treatment plan for non-invasive transcranial deep brain stimulation and verify safety.

DETAILED DESCRIPTION:
At present, those who are still ineffective after two or more full-dose antidepressants are called treatment-resistant depression (Treatment-Resistant Depression, TRD). Patients with TRD have increased suicide risk, increased medical expenditure, decreased quality of life, and increased disease burden. Existing diagnosis is verified by clinical symptoms, continuous attempts of antidepressant treatment programs, and observation of efficacy, lack of early identification of biological markers, and the main treatment strategies for TRD patients are related to side effects and high treatment resistance. Therefore, how to identify TRD early and intervene in time is an important direction of current depression research.

Based on the previous research work, this project plans to establish a prospective cohort study of clinical cases, and to discover the clinical characteristics of TRD, factors carried by peripheral blood and exosomes (Hypocretin, Brain-derived neurotrophic fact, Reelin, N-methyl-D- Aspartic acid receptor), functional magnetic resonance and brain electrophysiological indicators and other objective biological markers, using multi-modal fusion to establish an early identification model for TRD. At the same time, we plan to analyze the abnormal brain network characteristics and abnormal EEG phase characteristics of TRD, in order to search for abnormalities through multi-dimensional data Potential spatial and temporal intervention targets dependent on TRD status.

Recently, a new non-invasive transcranial electrical stimulation method, namely Temporal Interference Stimulation (TIS), can non-invasively stimulate area-specific Focus on the deep brain area without affecting the upper brain area of the target area. This project will carry out the research and development of the principle prototype of the non-invasive transcranial deep electric Clinical curative effect comparison and safety evaluation, so as to verify the best TIS intervention target, on this basis, according to the above-explored TRD state-dependent EEG signals, through spontaneous synchronous oscillation signals between different channels on the neural loop , to achieve individualized neuromodulation. Finally, a diagnosis and treatment model for early identification of refractory depression and non-invasive transcranial deep electrical stimulation technology will be established to provide new guidance for TRD treatment.

ELIGIBILITY:
Inclusion Criteria:

* This episode meets the diagnostic criteria of DSM-5 major depression, and is not accompanied by psychotic symptoms in the first episode or relapse of unmedicated depression;
* 24 item Hamilton Depression Scale (HAMD-24)≥20;
* Age 18-60, gender unlimited;
* right hand;
* Han Chinese;
* Sign a written informed consent and be willing to participate in the study and be evaluated.

Exclusion Criteria:

* Comorbidities with other mental disorders, including schizophrenia, mental retardation, substance dependence, etc.
* Patients with metal objects in the body or other contraindications for MRI scanning;
* Suffering from a serious or unstable physical disease;
* Positive urine HCG test results of pregnant and lactating women and women of childbearing age during screening;
* Other conditions deemed unsuitable for participation in the clinical trial by the investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 400 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Hamilton Depression Scale (24-items) Total Score Change | Baseline to end of stimulation period, an average of 14 days
  The Hamilton Depression Scale (24-items), is a 24 item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. It's considered the gold standard for rating depression severity and used frequently in clinical trials. Higher HAM-D24 score indicates more severe depression, and each item yields a score of 0 to 4. Remission is defined as HAM-D24 ≤8. A reduction of 50% or more in total score from Baseline indicates clinical response.

SECONDARY OUTCOMES:
Change of Hamilton Depression Scale (24-items) score | 7 days and 28 days
  The Hamilton Depression Scale (24-items), is a 24 item diagnostic questionnaire used to measure the severity of depressive episodes in patients with mood disorders. It's considered the gold standard for rating depression severity and used frequently in clinical trials. Higher HAM-D24 score indicates more severe depression, and each item yields a score of 0 to 4. Remission is defined as Change of Hamilton Depression Scale (24-items) ≤8. A reduction of 50% or more in total score from Baseline indicates clinical response.
Change in the rate of Beck Scale of Suicidal Ideation score | Baseline to end of stimulation period, an average of 14 days.
  Beck Scale of Suicidal Ideation is a 21-item self-report instrument that detects and measures the intensity of a patient's specific attitudes, behaviors, and suicide plans during the past week. The BSI score ranges from 0 to 63, with higher scores indicating worse outcomes and lower scores indicating better outcomes.
Change in the rate of Hamilton Anxiety Scale score | Baseline to end of stimulation period, an average of 14 days
  Hamilton Anxiety Scale is a 17 item diagnostic questionnaire used to measure the severity of anxiety episodes in patients. Each item on the scale is rated on a 5-point scale from 0 (not present) to 4 (severe), with the total score ranging from 0 to 68. The HAMA-17 is often used in clinical and research settings to assess the severity of anxiety symptoms and to evaluate the effectiveness of treatments for anxiety. It is a more comprehensive version of the HAMA that includes additional items to capture a broader range of anxiety symptoms.
Change in the score of THINC-it. | Baseline to end of stimulation period, an average of 14 days
  THINC-it is a computerized cognitive screening tool that is designed to assess cognitive function in adults. THINC-it stands for "THINking Clearly," and it includes a series of brief tests that evaluate several cognitive domains, including attention, working memory, executive function, and processing speed. The tool is administered on a tablet or computer, and it takes approximately 20 minutes to complete.
Treatment Emergent Symptom Scale | through study completion, an average of 14 days.
  The Treatment Emergent Symptom Scale (TESS) is a clinical tool that is used to monitor and evaluate the side effects or adverse events associated with various types of psychiatric treatments. The TESS includes a comprehensive list of symptoms that are commonly associated with psychiatric treatments, including medications for depression, anxiety, bipolar disorder, schizophrenia, and other mental health conditions. These symptoms may include physical symptoms, such as nausea, dizziness, or fatigue, as well as psychological symptoms, such as anxiety, irritability, or insomnia.During a clinical trial or other treatment study, patients are typically asked to complete the TESS at regular intervals to report any symptoms that they may be experiencing. The scores on the TESS can then be used to monitor the incidence and severity of side effects, to compare the side effect profiles of different treatments, and to assess the overall tolerability of different treatments.
Change in neuroimaging using functional magnetic resonance | Baseline, 14 days
  Scanning functional magnetic resonance. Functional magnetic resonance imaging (fMRI) is a neuroimaging technique that is used to measure changes in brain activity by detecting changes in blood flow. In the context of major depression, fMRI has been used to study changes in brain function that may be associated with the condition. Research using fMRI in major depression has shown that there are alterations in the activity of certain brain regions in people with the condition. Specifically, fMRI studies have identified changes in the activity of the prefrontal cortex, the amygdala, and the hippocampus in people with major depression. Overall, fMRI has provided valuable insights into the neural mechanisms underlying major depression, and may help to inform the development of new treatments for the condition.
Change in electroencephalogram | through study completion, an average of 14 days.
  Electroencephalogram is collected from 64 electrodes. EEG can be used to identify patterns of brain activity that are associated with the condition and to inform treatment decisions. EEG can be a useful tool for identifying patterns of brain activity that are associated with TRD and for guiding treatment decisions. Neurofeedback and TMS are two approaches that have shown promise in the treatment of TRD. several parameters are analyzed to identify patterns of brain activity that may be associated with the condition. These parameters include:
  Alpha power, Beta power, Theta power, Delta power, Coherence, and more.
Change of blood factor levels | Baseline, 14 days
  Factors carried by peripheral blood and exosomes(Hypocretin, Brain-derived neurotrophic fact, Reelin, N-methyl-D-aspartic acid receptor and so on).

CONTACTS AND LOCATIONS:
Overall Officials: Manli Huang, Professor, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital of Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No